CLINICAL TRIAL: NCT03165604
Title: The Effect of Information on Physical Fitness Measures and Training in Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MeirMc0017-17CTIL
Record Dates: First submitted 2017-04-18; First posted 2017-05-24 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Childhood Obesity
Keywords: Physical fitness; Exercise; Childhood Obesity; Information
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Subjects will be given the same drink (water) in different packaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight (Active Comparator): 30 normal weight children will receive 2 types of information: standard information and positive information regarding a water drink before physical exercise
  Interventions: Other: standard information; Other: positive information
- Over weight (Active Comparator): 30 over weight children will receive 2 types of information: standard information and positive information regarding a water drink before physical exercise
  Interventions: Other: standard information; Other: positive information

INTERVENTIONS:
Other: standard information — The participates will be given a standard information regarding the water drink before physical activity
Other: positive information — The participates will be given positive information (the drink will be presented as an "energy" drink) regarding the drink before physical activity

SUMMARY:
In the present study the investigators will examine the impact of varying information (positive compared to standard information) concerning a drink for improving physical fitness in overweight children.

DETAILED DESCRIPTION:
The present study will explore the short and medium term effects of receiving information concerning a drink (water) (positive compared to standard information) on the physical fitness in overweight children.

Study subjects will be 30 overweight children aged 6 to 13, new participates in a nutritional, behavioral sport program,The control group of 30 normal weight children.

The first stage of the study the investigators will examine the short-term influence of different types of information concerning water on subjects' fitness which will be measured by treadmill performance. First, the water will be presented to the participants children as an ordinary water while in the second case it will be presented as an "energy drink".

The second stage of the study will examine the impact of varying information on the subjects' sports participation/level of physical activity over a 6 week period of training, Study subjects will be 30 over-weight children aged 6 to 13, who participate in a nutritional, behavioral sport program. During this period, information on the type of drink will be changed every week. Children will be assessed in all training sessions and their level of activity will be monitored to examine whether the information on the drink led to a different exercise behavior.

The study hypothesis is that the use of these positive information will increase participants' fitness and levels of activity compared to standard information.

ELIGIBILITY:
Inclusion Criteria:

* Pre pubertal children
* Study group: BMI precentiles over 85 (overweight and obese children)
* Control group: BMI precentiles between 5-85 (normal weight children)

Exclusion Criteria:

* Children with organic Disease
* Competitive athlete

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Running time (seconds) | up to 6 weeks
  Overall running time during aerobic treadmill fitness test

SECONDARY OUTCOMES:
Maximal heart rate (beats/min) | up to 6 weeks
  Maximal heart rate during aerobic treadmill fitness test

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanti-Oren S, Birenbaum-Carmeli D, Eliakim A, Pantanowitz M, Nemet D. The effect of placebo on endurance capacity in normal weight children - a randomized trial. BMC Pediatr. 2019 Jan 10;19(1):15. doi: 10.1186/s12887-019-1394-x. PMID 30630461